CLINICAL TRIAL: NCT01350609
Title: Single Dose Study to Compare the Pharmacokinetics as Well as Safety and Tolerability of a Novel Fixed Dose Combination of Nifedipine GITS and Candesartan and the Loose Combination of Both Components and to Investigate the Bioequivalence Between the Fixed Dose and the Loose Combination in Healthy Male Subjects Under Fed Conditions in an Open Label, Randomized, 2-way-crossover Design
Brief Title: Pivotal Bioequivalence FDC Nifedipine / Candesartan vs. Loose Combination of Single Components, Fed
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 14028; 2011-000322-29 (EudraCT Number)
Record Dates: First submitted 2011-04-18; First posted 2011-05-10 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Hypertension, Essential
Keywords: essential hypertension, blood pressure, nifedipine, candesartan, FDC
MeSH Terms: conditions — Essential Hypertension | interventions — Nifedipine; candesartan; candesartan cilexetil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nifedipine/Candesartan (fixed dose) (Experimental)
  Interventions: Drug: Nifedipine/Candesartan (BAY 98-7106)
- Nifedipine/Candesartan (loose) (Active Comparator)
  Interventions: Drug: Nifedipine (Adalat, BAY A1040) and Candesartan (Atacand, BAY 12-9333)

INTERVENTIONS:
Drug: Nifedipine/Candesartan (BAY 98-7106) — Fixed dose combination of 60 mg nifedipine + 32 mg candesartan (1 tablet in one period)
  Arms: Nifedipine/Candesartan (fixed dose)
Drug: Nifedipine (Adalat, BAY A1040) and Candesartan (Atacand, BAY 12-9333) — Loose combination of 1 tablet nifedpipine 60mg (Adalat LA) and 2 tablets candesartan 16mg (Atacand) (3 tablets in one period) .
  Arms: Nifedipine/Candesartan (loose)

SUMMARY:
Randomized, open label, single dose, 2-way crossover study to investigate the bioequivalence of a new fixed dose combination (FDC) tablet of nifedipine GITS and candesartan with the corresponding loose combination under fed conditions.

DETAILED DESCRIPTION:
Clinical pharmacology

ELIGIBILITY:
Inclusion Criteria:

* The informed consent form must be signed before any study specific tests or procedures are done
* Confirmation of the subject's health insurance coverage prior to the first screening visit
* Healthy male subject
* Ethnicity: Caucasian
* Age: 18 to 45 years (inclusive) at the first screening visit
* Body mass index (BMI) above or equal 18, and below or equal 29.9 kg / m²
* Ability to understand and follow study-related instructions

Exclusion Criteria:

* Suspicion of drug or alcohol abuse
* Regular daily consumption of more than 1 L of xanthin-containing beverages
* Intake of foods or beverages containing grapefruit within 2 weeks prior to the first study drug administration (the same applies to pomelos and St. John's Wort)
* Use of medication within 4 weeks prior to the first study drug administration which could interfere with the investigational products (e.g. CYP3A inhibitors or CYP3A inducers)

  * examples for CYP3A inhibitors: erythromycin, inhibitors of human HIV protease (e.g. ritonavir, saquinavir), amiodarone, diltiazem, verapamil, fluconazole, itraconazole, ketoconazole, clarithromycin, telithromycin, nefazodon, cimetidine;
  * examples for CYP3A inducers: rifampicin, carbamazepin, phenytoin, phenobarbital, or products containing St. John's Wort;
* Systolic blood pressure below 116 or above 145 mmHg (after at least 15 min supine)
* At the first screening visit

  * Diastolic blood pressure above 95 mmHg (after at least 15 min supine)
  * Heart rate below 45 or above 95 beats / min (after at least 15 min supine) at the first screening visit
  * Clinically relevant findings in the physical examination
  * Positive urine drug screening or alcohol breath test
* Exclusion periods from other studies or simultaneous participation in other clinical studies

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2011-04; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Cmax | within 48 hours after each dosing
  Maximum drug concentration in plasma after dose administration for nifedipine and candesartan
AUC(0-tlast) | within 48 hours after each dosing
  Area under the drug-concentration vs. time curve from time 0 to the last data point for nifedipine and candesartan

SECONDARY OUTCOMES:
AUC | Within 48 hours after each dosing
  Area under the curve from time 0 to infinity after single dose for nifedipine and candesartan
Cmax,norm | Within 48 hours after each dosing
  Dose normalized Cmax for nifedipine and candesartan
AUCnorm | Within 48 hours after each dosing
  AUC normalized for dose and body weight for nifedipine and candesartan
AUC(0-48) | Within 48 hours after each dosing
  Area under the plasma concentration-time curve from time zero to 48h for nifedipine and candesartan
Tmax | Within 48 hours after each dosing
  The time of the maximum concentration for nifedipine and candesartan
t1/2 | Within 48 hours after each dosing
  Half-life for nifedipine and candesartan
MRT | Within 48 hours after each dosing
  The mean residence time for nifedipine and candesartan
CL/F | Within 48 hours after each dosing
  Oral plasma clearances for nifedipine and candesartan
Number of participants with adverse events | Approximately 3-7 weeks per subject

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Berlin, State of Berlin, Germany

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/